CLINICAL TRIAL: NCT01757782
Title: Oral Sildenafil in Persistent Pulmonary Hypertension of Neonates Secondary to Meconium Aspiration Syndrome: A Randomized Placebo Controlled Trial
Brief Title: Oral Sildenafil in Persistent Pulmonary Hypertension Secondary to Meconium Aspiration Syndrome in Newborns
Acronym: OSiNPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Takhtasinhji General Hospital (Other Government)
Responsible Party: Principal Investigator, Jayendra R. Gohil, MD, PROF., Professor in Pediatrics, Sir Takhtasinhji General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sildenafil
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Meconium Aspiration Syndrome; Persistent Pulmonary Hypertension of Newborn
Keywords: MAS; PPHN; Sildenafil; Newborn; Pulmonary Hypertension
MeSH Terms: conditions — Meconium Aspiration Syndrome; Persistent Fetal Circulation Syndrome; Hypertension, Pulmonary | interventions — Sildenafil Citrate; integra artificial skin; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Sildenafil (Active Comparator): In group A, newborns received oral Sildenafil solution through feeding tube which was prepared by crushing a 50 mg tablet of sildenafil in distilled water to make a concentration of 5 mg/ml. The protocol for dosing was (1) first dose of 1 mg/kg/dose within 30 minutes admission or within 12 hours of delivery (whichever earlier), (2) Dosing every six hours for a maximum of 8 doses.
  Interventions: Drug: Oral Sildenafil
- Distilled water (Placebo Comparator): In group B, newborns received placebo. The protocol for dosing was (1) first dose of 1 mg/kg/dose within 30 minutes admission or within 12 hours of delivery (whichever earlier), (2) Dosing every six hours for a maximum of 8 doses.
  Interventions: Drug: Placebo (distilled water)

INTERVENTIONS:
Drug: Oral Sildenafil — Patients were randomized into two groups. Placebo was prepared with distilled water. In group A, newborns received oral Sildenafil solution through feeding tube which was prepared by crushing a 50 mg tablet of sildenafil in distilled water to make a concentration of 5 mg/ml. In group B, newborns received placebo. The protocol for dosing was (1) first dose of 1 mg/kg/dose within 30 minutes admission or within 12 hours of delivery (whichever earlier), (2) Dosing every six hours for a maximum of 8 doses, (3) Dose was doubled if the oxygenation index (OI) or SpO2 did not improve (If OI continued to be <10% of previous value and SpO2 was not increasing >5 of previous value) and blood pressure remained stable
  Other Names: Viagra; Integra
  Arms: Oral Sildenafil
Drug: Placebo (distilled water) — Distill water oral
  Other Names: Water
  Arms: Distilled water

SUMMARY:
The purpose of this study is to to study the role of oral Sildenafil in Persistent Pulmonary Hypertension of Newborn (PPHN) secondary to Meconium Aspiration Syndrome (MAS) in newborns and to study risk factors of MAS developing into PPHN.

DETAILED DESCRIPTION:
Design: Randomized control trial Setting: Neonatal intensive care unit in a tertiary care hospital Patients: Patients diagnosed with MAS with PPHN according to clinical criteria. 97 patients with MAS were enrolled in the study over a period of 8 months, out of which 40 patients with PPHN were randomized into two groups.

Intervention: Group A received Sildenafil through a feeding tube (1 mg/kg/dose q6h) for 8 doses. Group B received a placebo. Outcome measures: Improvement in oxygen saturation (SpO2), oxygenation index (OI), duration of hospitalization and mechanical ventilation and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Newborns were diagnosed with MAS if any of the two of the following three criteria were present. (1) Meconium staining of liquor or staining of umbilical cord or skin or nails. (2) Respiratory distress, within one hour of birth. (3) Radiological evidence of aspiration pneumonitis (atelectasis and/or hyperinflation). Newborns with MAS diagnosed with clinical PPHN were enrolled in the study for drug trial. PPHN was determined either clinically by loud P2(second component of second heart sound), 10% or greater pre-/post ductal difference in arterial oxygenation (obtained by acid base gas analysis) or upper limb- lower limb SpO2 difference (obtained by pulse oximetry).

Exclusion Criteria:

* (a) babies with congenital heart disease (b) congenital anomalies particularly those which were incompatible to life or which was the cause for respiratory distress e.g. diaphragmatic hernia (c) Respiratory morbidities such as hyaline membrane disease, congenital pneumonia (d) Babies with PPHN secondary to MAS admitted after 12 hours of delivery (e) Non availability of consent of guardian for interventional procedures

Ages: 1 Minute to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Improvement in oxygen saturation (SpO2) | 26 hours, 50 hours
  Preductal and postductal oxygen saturation (SpO2) 2 hours after dose of oral sildenafil (24 hours and 48 hours)

SECONDARY OUTCOMES:
Oxygenation index | 26 hours, 50 hours
  Oxygenation index of neonates kept on ventilator 2 hours after dose of oral sildenafil (24 hours and 48 hours) [Oxygenation index (OI) = Mean airway pressure (cm H2O) × FiO2 × 100/ PaO2 [fraction of inspired oxygen- FiO2] [Arterial partial pressure of oxygen- PaO2]

OTHER OUTCOMES:
Mortality of patients enrolled in study | Upto 4 weeks
  During time of hospital stay(upto 4 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Jayendra R Gohil, MD, Principal Investigator — Professor Pediatrics, Govt Medical College, Bhavnagar, Gujarat, India
Locations (1):
- NICU, Pediatrics department, SirTakhtasinhjiGH, Bhavnagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: Yes
Available for six months on request
Supporting Information: CSR
Time Frame: six months
Access Criteria: on demand

REFERENCES:
- [Background] Vargas-Origel A, Gomez-Rodriguez G, Aldana-Valenzuela C, Vela-Huerta MM, Alarcon-Santos SB, Amador-Licona N. The use of sildenafil in persistent pulmonary hypertension of the newborn. Am J Perinatol. 2010 Mar;27(3):225-30. doi: 10.1055/s-0029-1239496. Epub 2009 Oct 28. PMID 19866403